CLINICAL TRIAL: NCT01873937
Title: COMPARATIVE CLINICAL STUDY OF LIGHT ANALGESIC EFFECT ON TEMPOROMANDIBULAR DISORDER (TMD) USING RED AND INFRARED LED-THERAPY
Brief Title: Analgesic Effects of LED Light on Temporomandibular Disorders.
Acronym: LED/TMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Fernanda Rossi Paolillo, Vitor Hugo Panhóca, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1967
Record Dates: First submitted 2013-05-29; First posted 2013-06-10 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Temporomandibular Disorder
Keywords: Lasertherapy; Ledtherapy; TMJs; pain relief; oral aperture
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Red LED (Experimental): Irradiation parameters: 630 nm, 60 sec and 18 J/cm² per point.
  Interventions: Radiation: Red LED
- infrared LED (Experimental): Irradiation parameters: 850 nm, 60 sec and 18J/cm² per point
  Interventions: Radiation: INFRARED LED
- LASER (Active Comparator): Irradiation parameters: 780 nm, 60 sec and 105 J/cm²
  Interventions: Radiation: LASER

INTERVENTIONS:
Radiation: Red LED — Phototherapy with red LED on temporomandibular area
  Other Names: Irradiation parameters: 630 nm, 60 sec and 18 J/cm² per point.
  Arms: Red LED
Radiation: INFRARED LED — Phototherapy with infrared LED on temporomandibular area
  Other Names: Irradiation parameters: 850 nm, 60 sec and 18J/cm² per point
  Arms: infrared LED
Radiation: LASER — Phototherapy with LASER INFRARED on temporomandibular area
  Other Names: Irradiation parameters: 780 nm, 60 sec and 105 J/cm²
  Arms: LASER

SUMMARY:
Low intensity laser therapy (LILT) has been widely applied in pain relief in several clinical situations. With the advent of new LED-based (light emitting diode) light sources, the need of further clinical experiments aiming to compare the effectiveness between them is paramount.

DETAILED DESCRIPTION:
Aims: Low intensity laser therapy (LILT) has been widely applied in pain relief in several clinical situations. With the advent of new LED-based (light emitting diode)light sources, the need of further clinical experiments aiming to compare the effectiveness between them is paramount. Method: This study proposes an evaluation of analgesic effect in TMD (temporomandibular disorders) using two different LEDs systems, one emitting at the spectral band of red (630 +/-5 nm) and the other at infrared band (850 +/-5 nm), and compare the results with a laser treated control group (780nm diode laser using 105.7 J/cm2). Mandibular range of motion and report of pain were evaluated via appropriate equipment developed to do this end. Power output was 150mW, tip area was 0.5 cm² for both sources. Fluency or dose chosen was 18 J/cm² for each point of application, around the TMJ, on both sides. Five points were irradiated on TMJ, temporal and masseter muscles. Eight irradiation sessions were done and follow up was performed 7 and 30 days, after last session. Thirty patients were enrolled and they were selected randomly for each treatment, resulting in 10 patients per group (infrared LED, red LED and Control Group using infrared Laser).

ELIGIBILITY:
Inclusion Criteria:

Thirty patients (from 18 to 50 years old) presenting signs and symptoms of TMD were selected to participate in the study. The patients received care at a private dental office in Ribeirao Preto, São Paulo, Brazil (NILO- Integrated Center for Laser in Dentistry). The patients´ age ranged from 18 to 40 years old, being 08 male and 22 female. The signs and symptoms evaluated by a trained professional were as follow: pain during palpation in the TMJ area, pain on associated muscles (masseter and temporal), and limited or painful jaw movement with impaired oral aperture.

Exclusion Criteria:

The exclusion criteria were patients whom where currently under orthodontic and/or orthopedic treatment, degenerative joint disease, patients who were under systemic medication with anti-inflammatory drugs, analgesic treatment, muscle relaxant and corticosteroids.

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Relationships between pain and range of motion | 2 months
  Pain score and mandibular range of motion

SECONDARY OUTCOMES:
Research Diagnostic Criteria(RDC)/Temporomandibular Disorders (DTM) | 2 months
  RDC/DTM diagnostic exam for research of arthralgia and chronic myofascial pain. The signs and symptoms evaluated by a trained professional were as follow: pain during palpation in the temporomandibular joint, pain on associated muscles (masseter and temporal), and limited or painful jaw movement with impaired oral aperture.

CONTACTS AND LOCATIONS:
Overall Officials: Panhóca H Panhóca, MS, Principal Investigator — IFSC/UFSCAR; Rosane Z Lizarelli, PhD, Study Director — University of São Paulo, IFSC; Vanderlei S Bagnato, PhD, Study Director — University of São Paulo, IFSC
Locations (1):
- NILO- Integrated Center for Laser in Dentistry, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Result] Vinck E, Coorevits P, Cagnie B, De Muynck M, Vanderstraeten G, Cambier D. Evidence of changes in sural nerve conduction mediated by light emitting diode irradiation. Lasers Med Sci. 2005;20(1):35-40. doi: 10.1007/s10103-005-0333-2. Epub 2005 May 14. PMID 15895289
- [Result] Whelan HT, Connelly JF, Hodgson BD, Barbeau L, Post AC, Bullard G, Buchmann EV, Kane M, Whelan NT, Warwick A, Margolis D. NASA light-emitting diodes for the prevention of oral mucositis in pediatric bone marrow transplant patients. J Clin Laser Med Surg. 2002 Dec;20(6):319-24. doi: 10.1089/104454702320901107. PMID 12513918
- [Result] Hansson TL. Infrared laser in the treatment of craniomandibular disorders, arthrogenous pain. J Prosthet Dent. 1989 May;61(5):614-7. doi: 10.1016/0022-3913(89)90287-4. PMID 2746531
- [Result] Oz S, Gokcen-Rohlig B, Saruhanoglu A, Tuncer EB. Management of myofascial pain: low-level laser therapy versus occlusal splints. J Craniofac Surg. 2010 Nov;21(6):1722-8. doi: 10.1097/SCS.0b013e3181f3c76c. PMID 21119408
- See also: Related Info — http://cepof.ifsc.usp.br/